CLINICAL TRIAL: NCT02525770
Title: Comparative Study of the Wear of Uncemented Acetabular Conventional Polyethylene and X3 in Total Hip Replacement, for Stereo-radiographic Analysis
Acronym: COCYCOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-018
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Radiostereometric Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acetabular liner in X3 polyethylene (Active Comparator): acetabular in X3 polyethylene
  Interventions: Device: radiostereometric analysis (RSA)
- acetabular liner in N2VAC® conventional polyethylene (Active Comparator): hip replacement with acetabular liner in N2VAC® conventional polyethylene
  Interventions: Device: radiostereometric analysis (RSA)

INTERVENTIONS:
Device: radiostereometric analysis (RSA)

SUMMARY:
Total hip arthroplasty (THA) is one of the most effective medical procedures. Except for the few early complications (acute infections and dislocations), the patient made a PTH can be assured of a significant improvement in its function and its short-term quality of life. However, clinical studies and records have shown that the lifetime of these implants was limited. The main cause of failure is the "aseptic loosening" influenced by many factors, foremost of which is due to periprosthetic osteolysis debris. This is a major concern for orthopedic surgeons loosening leads, in most cases, the recovery, the importance of osteolysis is a major cause of difficulties and poorer results.

The main objective of the study is to compare, 2 years after the intervention, the penetration of the femoral head in the polyethylene and X3 in the acetabulum in N2VAC® conventional polyethylene.

ELIGIBILITY:
Inclusion Criteria:

* Patient (18-70 years) with hip disease necessitating the establishment of a total hip replacement

Exclusion Criteria:

* Patient aged 71 or more
* Pregnant woman or wishing to be for the duration of the study
* Resumption of total hip replacement, or cephalic prosthesis cups
* Primary or secondary malignant neoplasm of the hip
* Protected adult patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2010-06; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Penetration of the femoral head in the polyethylene measure in millimeters | change over baseline and 2 years
  The median head penetration in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'orthopédie traumatologie, CHu de Caen, Caen, France